CLINICAL TRIAL: NCT02202915
Title: CBT for Pediatric OCD: Community Training Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Kristen Benito, Ph.D., Assistant Professor/Staff Psychologist, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4R33MH096828-03 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fidelity Checklist Arm (Experimental): Therapists are receiving training using the fidelity Checklist
  Interventions: Behavioral: Behavioral Checklist

INTERVENTIONS:
Behavioral: Behavioral Checklist

SUMMARY:
This study examines a training program for clinicians who work in mental health clinics that serve children with OCD. We will provide clinician training in conducting exposure-based treatments for children with OCD. The purpose of the project is to test the use of a new tool to enhance training in exposure-based treatments for clinicians. Therapists will receive training and oversight from the researchers regarding the treatment procedures and use of the new tool. All children enrolled in the study will receive treatment by clinicians who are participating in this study. Therapists and youth will be recruited separately for the study and will be assigned to work together.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive Compulsive Disorder is primary diagnosis

Exclusion Criteria:

* Diagnosis of Psychosis, Pervasive Developmental Disorder, or Mental Retardation

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Observed therapist behaviors | 9 months
  We will us the Exposure Process Coding System to identify behaviors that therapists used during the exposures

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley Hospital, East Providence, Rhode Island, United States